CLINICAL TRIAL: NCT00437268
Title: A Randomized Phase 2 Study of Irinotecan Plus Cetuximab With or Without Enzastaurin in Patients With Recurrent Colorectal Cancer
Brief Title: A Study of Irinotecan Plus Cetuximab With or Without Enzastaurin in Participants With Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10538; H6Q-MC-S018 (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-02-16; First posted 2007-02-19 (Estimated); Results first posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Colorectal Cancer; Colorectal Carcinoma; Colorectal Tumor
MeSH Terms: conditions — Colorectal Neoplasms | interventions — enzastaurin; Irinotecan; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- enzastaurin + irinotecan + cetuximab (Experimental)
  Interventions: Drug: enzastaurin; Drug: irinotecan; Drug: cetuximab
- irinotecan + cetuximab (Active Comparator)
  Interventions: Drug: irinotecan; Drug: cetuximab

INTERVENTIONS:
Drug: enzastaurin — 1125 milligrams (mg) loading dose, then 500 mg orally, daily, of each 21-day cycle until progressive disease
  Other Names: LY317615
  Arms: enzastaurin + irinotecan + cetuximab
Drug: irinotecan — 300 milligrams per square meter (mg/m^2) intravenously on Day 1 of each 21-day cycle until progressive disease
Drug: cetuximab — 400 mg/m^2, intravenously on Day 1, 250 mg/m^2 on Day 8, Day 15 Cycle 1 then 250 mg/m^2, on Day 1, 8 and 15 of each cycle, intravenously 21-day cycles until progressive disease

SUMMARY:
To see how well enzastaurin in combination with irinotecan and cetuximab works versus irinotecan and cetuximab in participants who have progressed within 3 months.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if they meet all of the following criteria:

1. Histologic diagnosis of colorectal cancer.
2. Performance status of 0, 1, or 2 on the Eastern Cooperative Oncology Group (ECOG) performance status schedule.
3. Have had documented disease progression according to Response Evaluation Criteria in Solid Tumors (RECIST v1.0; Therasse et al. 2000) within 3 months after receiving 5-fluorouracil, leucovorin, and oxaliplatin (FOLFOX) plus bevacizumab as first-line therapy for locally advanced or metastatic disease, or within 6 months after receiving FOLFOX with or without bevacizumab in the adjuvant setting.
4. Standard radiation therapy for rectal cancer is allowed. Participants must have recovered from the toxic effects (except for alopecia) of the treatment prior to study enrollment. Prior radiotherapy must be completed 4 weeks before study entry. Lesions that have been radiated in the advanced setting cannot be included as sites of measurable disease unless clear tumor progression has been documented in these lesions since the end of radiation therapy.
5. At least one uni-dimensionally measurable lesion meeting RECIST v1.0 guidelines (at least 10 millimeters [mm] in longest diameter by spiral computerized tomography (CT) scan, or at least 20 mm by standard techniques). Positron emission tomography (PET) scans and ultrasounds may not be used.

Exclusion Criteria:

Participants will be excluded from the study if they meet any of the following criteria:

1. Have received treatment within the last 4 weeks with a drug that has not received regulatory approval for any indication at the time of study entry.
2. Have previously completed or withdrawn from this study or any other study investigating enzastaurin, irinotecan, or cetuximab.
3. Have a serious concomitant systemic disorder [such as active infection including human immunodeficiency virus (HIV), or cardiac disease] that, in the opinion of the investigator, would compromise the participant's ability to adhere to the protocol.
4. Have a serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease, as defined by the New York Heart Association Class III or IV.
5. Have a prior malignancy (other than colorectal cancer, or adequately treated carcinoma in-situ of the cervix or nonmelanoma skin cancer), unless that prior malignancy was diagnosed and definitively treated at least 5 years previously with no subsequent evidence of recurrence. Participants with a history of low grade (Gleason score less than or equal to 6) localized prostate cancer will be eligible even if diagnosed less than 5 years previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-03; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours,EST), Study Director — Eli Lilly and Company
Locations (20):
- United States (20):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Casa Grande, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tucson, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Springs, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orlando, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington Heights, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shreveport, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kalamazoo, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Robbinsdale, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valhalla, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Worth, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubbock, Texas

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant flow reports those participants who discontinued from study drug.
Groups:
- Enzastaurin+Irinotecan+Cetuximab: Enzastaurin: 1125 milligrams (mg) loading dose on Day 1 of Cycle 1, then 500 mg orally, daily, of each 21-day cycle until progressive disease
  Irinotecan: 300 milligrams per square meter (mg/m^2), intravenously on Day 1 of each 21-day cycle until progressive disease
  Cetuximab: 400 mg/m^2 intravenously on Day 1, then 250 mg/m^2 on Days 8 and 15 of Cycle 1, then 250 mg/m^2 on Days 8 and 15 in Cycle 1, then 250 mg/m^2 intravenously on Days 1, 8 and 15 of each 21-day cycle until progressive disease
- Irinotecan+Cetuximab: Irinotecan: 300 mg/m^2 intravenously on Day 1 of each 21-day cycle until progressive disease
  Cetuximab: 400 mg/m^2 intravenously on Day 1, then 250 mg/m^2 on Days 8 and 15 in Cycle 1, then 250 mg/m^2 intravenously on Days 1, 8 and 15 of each 21-day cycle until progressive disease
Period: Overall Study
Arm/Group | Enzastaurin+Irinotecan+Cetuximab | Irinotecan+Cetuximab
Started | 13 | 13
Received at Least 1 Dose of Study Drug | 13 | 13
Protocol Qualified (PQ) Participant | 13 (PQ population: randomized participants without an immune reaction to cetuximab after the first dose) | 12 (PQ population: randomized participants without an immune reaction to cetuximab after the first dose)
Completed | 0 | 0
Not Completed | 13 | 13
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Progressive disease | 9 | 9
Not completed — Physician Decision | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Enzastaurin+Irinotecan+Cetuximab: Enzastaurin: 1125 milligrams (mg) loading dose on Day 1 of Cycle 1, then 500 mg orally, daily, of each 21-day cycle until progressive disease
  Irinotecan: 300 mg/m^2 intravenously on Day 1 of each 21-day cycle until progressive disease
  Cetuximab: 400 mg/m^2 intravenously on Day 1, then 250 mg/m^2 on Days 8 and 15 in Cycle 1, then 250 mg/m^2 intravenously on Days 1, 8 and 15 of each 21-day cycle until progressive disease
- Total: Total of all reporting groups
Arm/Group | Enzastaurin+Irinotecan+Cetuximab | Irinotecan+Cetuximab | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.5 (12.45) | 59.5 (10.28) | 56.0 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 9 | 10 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5 | 10 | 15
  Black or African American | 2 | 0 | 2
  Asian | 2 | 0 | 2
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 13 | 26
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status classifies participants according to their functional impairment.
  Participants
    0 - Fully Active | 4 | 6 | 10
    1 - Ambulatory, Restricted Strenuous Activity | 9 | 7 | 16
Adjuvant Therapy Status [Count of Participants; unit: Participants]
  Yes | 7 | 5 | 12
  No | 6 | 8 | 14
Basis for Initial Diagnosis [Count of Participants; unit: Participants]
  Histopathologic | 10 | 13 | 23
  Cytologic | 3 | 0 | 3
Stage of Disease at Initial Diagnosis [Count of Participants; unit: Participants] — Cancer staging is a process describing the severity of the cancer, size of the tumor, and how far it has spread from the original location.
  Stage IIb - invaded adjacent organs or penetrates peritoneum (outer lining of the colon); Stage IIIb - has spread to 1-3 nearby nodes; Stage IIIc - has spread to ≥ 4 nearby nodes; Stage IV - the cancer has spread to other organs of the body such as the lung, brain, or liver.
  Participants
    Stage IIB | 1 | 0 | 1
    Stage IIIB | 1 | 0 | 1
    Stage IIIC | 0 | 2 | 2
    Stage IV | 11 | 11 | 22
Disease Type at Initial Diagnosis [Count of Participants; unit: Participants]
  Adenocarcinoma | 12 | 10 | 22
  Mucinous Adenocarcinoma | 1 | 2 | 3
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-Free Survival (PFS) at 6 Months (PFS Rate)
Description: PFS was defined as the time from the date of study enrollment to the first date of progressive disease or death from any cause. For participants not known to have died as of the data cut-off date and who did not have progressive disease, PFS was censored at the date of last visit with adequate assessment. For participants who received subsequent anticancer therapy (after discontinuation from the study treatment) prior to disease progression or death, PFS was censored at the date of last visit with adequate assessment prior to the initiation of post-discontinuation anticancer therapy. The PFS probability values were multiplied by 100 to obtain the percentage values.
Time Frame: At 6 months from randomization
Population: Protocol qualified population: All randomized participants who received at least 1 dose of study drug and did not develop a severe infusion reaction to cetuximab after the first dose. Participants censored: Irinotecan +Cetuximab+Enzastaurin = 1; Irinotecan +Cetuximab =2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin+Irinotecan+Cetuximab | Irinotecan+Cetuximab
Number analyzed (Participants) | 13 | 12
percentage of participants | 26 [1 to 51] | 23 [0 to 49]
Statistical Analysis 1: Comparison: Enzastaurin+Irinotecan+Cetuximab vs Irinotecan+Cetuximab; Test type: Superiority or Other; p = 0.431, Log Rank — The type 1 error rate was set at 0.20

2. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) (Tumor Response Rate)
Description: Tumor response rate was defined as number of participants with overall best response of complete response (CR) or partial response (PR) over number of protocol qualified participants using the Response Evaluation Criteria in Solid Tumors (RECIST v1.0) Guidelines. CR was defined as the disappearance of all tumor lesions. PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum of LDs or complete disappearance of target lesions, with persistence (but not worsening) of 1 or more non-target lesions, with no new lesions appearing. Percentage of participants = (Number of participants with overall best response of CR or PR/Number of protocol qualified participants) x 100.
Time Frame: Baseline to measured progressive disease up to 13.2 months
Population: Protocol qualified population: All randomized participants who received at least 1 dose of study drug and did not develop a severe infusion reaction to cetuximab after the first dose.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Irinotecan+Cetuximab: Irinotecan: 300 milligrams per square meter (mg/m^2), intravenously on Day 1 of each 21-day cycle until progressive disease
  Cetuximab: 400 mg/m^2 intravenously on Day 1, then 250 mg/m^2 on Days 8 and 15 of Cycle 1, then 250 mg/m^2 intravenously on Days 1, 8 and 15 of each 21-day cycle until progressive disease
Arm/Group | Enzastaurin+Irinotecan+Cetuximab | Irinotecan+Cetuximab
Number analyzed (Participants) | 13 | 12
percentage of participants | 7.7 [0.2 to 36.0] | 16.7 [2.1 to 48.4]
Statistical Analysis 1: Comparison: Enzastaurin+Irinotecan+Cetuximab vs Irinotecan+Cetuximab; Test type: Superiority or Other; p = 0.593, Fisher Exact

3. Secondary Outcome: Duration of Response
Description: The duration of a complete response (CR) or partial response (PR) was defined as the time from first objective status assessment of CR or PR to the first time of disease progression or death from any cause. According to the Response Evaluation Criteria in Solid Tumors (RECIST v1.0) criteria, CR was defined as the disappearance of all tumor lesions and PR was defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions taking as reference the baseline sum of LDs or complete disappearance of target lesions, with persistence (but not worsening) of 1 or more non-target lesions, with no new lesions appearing. For participants who died, the duration of response was censored at death. For participants still alive, duration of response was censored at the last visit with adequate assessment.
Time Frame: Time of response to progressive disease up to 13.2 months
Population: Participants with a CR or PR. No participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Enzastaurin+Irinotecan+Cetuximab: Enzastaurin: 1125 milligrams (mg) loading dose on Day 1 of Cycle 1, then 500 mg orally, daily, of each 21-day cycle until progressive disease
  Irinotecan: 300 milligrams per square meter (mg/m^2), intravenously on Day 1 of each 21-day cycle until progressive disease
  Cetuximab: 400 mg/m^2 intravenously on Day 1, then 250 mg/m^2 on Days 8 and 15 of Cycle 1, then 250 mg/m^2 intravenously on Days 1, 8 and 15 of each 21-day cycle until progressive disease
Arm/Group | Enzastaurin+Irinotecan+Cetuximab | Irinotecan+Cetuximab
Number analyzed (Participants) | 1 | 2
months | 6.9 [NA to NA] — The confidence interval was not estimable due to too few data points | 12.6 [12.0 to 13.2]
Statistical Analysis 1: Comparison: Enzastaurin+Irinotecan+Cetuximab vs Irinotecan+Cetuximab; Test type: Superiority or Other; p = 0.157, Log Rank

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time in months from the date of study enrollment to the date of death from any cause. For participants not known to have died as of the cut-off date, OS was censored at the last contact date.
Time Frame: Randomization to date of death from any cause up to 21.9 months
Population: Protocol qualified population: All randomized participants who received at least 1 dose of study drug and did not develop a severe infusion reaction to cetuximab after the first dose. Censored participants: Enzastaurin+Irinotecan+Cetuximab = 4; Irinotecan+Cetuximab = 4.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Enzastaurin+Irinotecan+Cetuximab | Irinotecan+Cetuximab
Number analyzed (Participants) | 13 | 12
months | 8.5 [5.5 to 16.4] | 8.0 [4.5 to 21.9]
Statistical Analysis 1: Comparison: Enzastaurin+Irinotecan+Cetuximab vs Irinotecan+Cetuximab; Test type: Superiority or Other; p = 0.539, Log Rank — Kaplan-Meier analysis was used for statistical analysis

5. Secondary Outcome: Percentage of Participants With a Complete Response (CR), Partial Response (PR) or Stable Disease (SD) (Disease Control Rate)
Description: The overall disease control rate for each treatment arm was calculated as percent of participants with overall response of complete response (CR), partial response (PR) or stable disease (SD) over number of protocol qualified population. According to the Response Evaluation Criteria in Solid Tumors (RECIST v1.0) criteria, CR was defined as the disappearance of all tumor lesions, PR was defined as at least a 30% decrease in sum of longest diameter (LD) of target lesions, progressive disease (PD) was defined as at least 20% increase in sum of LD of target lesions, and SD was defined as small changes that did not meet above criteria.
  Percentage of participants = (Number of participants with overall best response of CR, PR, or SD/Number of protocol qualified participants) x 100.
Time Frame: Baseline to disease progression (up to 13.2 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzastaurin+Irinotecan+Cetuximab | Irinotecan+Cetuximab
Number analyzed (Participants) | 13 | 12
percentage of participants | 38.5 [13.9 to 68.4] | 50.0 [21.1 to 78.9]
Statistical Analysis 1: Comparison: Enzastaurin+Irinotecan+Cetuximab vs Irinotecan+Cetuximab; Test type: Superiority or Other; p = 0.695, Fisher Exact

6. Secondary Outcome: Number of Participants With Adverse Events (AEs) or Who Died
Description: Clinically significant events were defined as serious and other non-serious AEs. Participants who died due to progressive disease (PD) or and adverse events (AEs) while on treatment and or died during the 30 day post-treatment are included. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline to study completion (Cycle 31.5 [21 days/cycle] and 30-day safety follow-up)
Population: The safety population included all randomized and treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzastaurin+Irinotecan+Cetuximab | Irinotecan+Cetuximab
Number analyzed (Participants) | 13 | 13
Participants
  Non-serious AEs | 13 | 13
  Serious AEs | 8 | 6
  Deaths Due to PD | 0 | 0
  Deaths Due to AEs | 0 | 1
  Deaths in 30-day follow-up | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline to study completion (Cycle 31.5 [21 days/cycle] and 30-day safety follow-up)
Description: Study-specific clinical outcomes due to progressive disease were not considered to be a serious adverse event (SAE) unless the investigator deemed it related to the use of the study drug.
Arm/Group | Enzastaurin+Irinotecan+Cetuximab | Irinotecan+Cetuximab
Serious Adverse Events (participants affected / at risk) | 8/13 | 6/13
Other Adverse Events (participants affected / at risk) | 13/13 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Enzastaurin+Irinotecan+Cetuximab (N=13) | Irinotecan+Cetuximab (N=13)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Gallbladder obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anorectal cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/9 (1) | 1/9 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzastaurin+Irinotecan+Cetuximab (N=13) | Irinotecan+Cetuximab (N=13)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (6)
Neutropenia (Blood and lymphatic system disorders) | 5 (7) | 5 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (4) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Erythema of eyelid (Eye disorders) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 6 (6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Breath odour (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (8) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 8 (11) | 9 (18)
Dry mouth (Gastrointestinal disorders) | 4 (5) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (10) | 11 (20)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (5) | 6 (7)
Asthenia (General disorders) | 1 (1) | 3 (4)
Chills (General disorders) | 1 (1) | 1 (1)
Cyst (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 8 (9) | 9 (13)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (2) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Xerosis (General disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Blood urea increased (Investigations) | 1 (1) | 0 (0)
Carcinoembryonic antigen increased (Investigations) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 2 (2)
Weight increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (3) | 4 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Oral neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 5 (5) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Chromaturia (Renal and urinary disorders) | 3 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6 (7) | 7 (7)
Drug eruption (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 5 (9) | 5 (6)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Results from other studies showed participants with mutant K-RAS tumors did not respond to Cetuximab. Due to issues with confounding of results the decision was to stop the study early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days